CLINICAL TRIAL: NCT05721482
Title: Addressing the Double Jeopardy of Stress and Hypertension Among African American Female Caregivers of Persons Living With Alzheimer's Disease and Related Dementias
Brief Title: Stress and Hypertension in Dementia Caregivers
Acronym: MIM-DASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kathy D. Wright, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2022B0031; R21AG077069 (NIH)
Record Dates: First submitted 2022-11-10; First posted 2023-02-10 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Stress, Psychological
Keywords: Dementia Caregivers
MeSH Terms: conditions — Hypertension; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized control trial of behavioral intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIM-DASH (Experimental): A trained MIM provider and dietitian will deliver the MIM DASH group intervention in eight weekly 1-hour sessions via telehealth.
  Interventions: Behavioral: Caregiver Training
- Attention Control (No Intervention): A trained interventionist will deliver the Caregiver Training. Participants in this group will attend eight 1-hour group lessons via telehealth for 8 weeks. We will use Alzheimer's Association caregiver training resources on topics such as Healthy Living for Your Brain and Body: Tips from the Latest Research; Dementia Conversations: Driving, Doctors Visits, Legal and Financial Planning; and Understanding and Responding to Dementia-Related Behavior. Similar to the MIM DASH group, participants will receive educational materials so they can follow along using videoconferencing or phone.

INTERVENTIONS:
Behavioral: Caregiver Training — A trained MIM provider and dietitian will deliver the MIM DASH group intervention in eight weekly 1-hour sessions via telehealth. Participants will receive session materials so they can follow along. Each MIM session consists of material related to mindfulness-the somatic mind/body connection, relaxation, yoga, meditation, self-awareness, and bodily cues relating to emotional reactivity. Group interaction centers on sharing ideas toward effective practice and practical daily challenges to being mindful. Each class begins with a prompt for participant contemplation during the next hour that reference a unique weekly theme which will be reiterated in the session materials.
  The DASH portion, led by the Registered Dietitian, focuses on education to increase vegetables, fruits, whole grains and decrease intakes of fat and sodium, sugar sweetened beverages and sweets. Education includes adapting traditional "Soul" food dishes to meet the DASH dietary guidelines.
  Other Names: MIM-DASH
  Arms: MIM-DASH

SUMMARY:
No demographic group is more at risk for the double jeopardy of caregiving stress and hypertension (HTN) than African American women caring for a family member with Alzheimer's disease and related dementias (ADRD). Both situations lead to reduced quality of life and cardiovascular disease-a complication of uncontrolled hypertension. Maintaining the health of these caregivers is critical to support the well-being of the care recipients. Although some multi-component interventions have addressed ADRD caregiver's stress and quality of life, gaps remain in targeting interventions to address the complexity of chronic caregiving stress and hypertension self-care in African American women.

This pilot study builds on the investigator's earlier work which showed that stress, blood pressure knowledge, and complex diet information deficits all interfered with older African American women's hypertension self-care. Lifestyle changes (stress management, reducing sodium, eating fruits/vegetables, and physical activity) are effective in managing hypertension. The investigator's Stage I pilot study is based on the scientific rationale that these lifestyle changes can be promoted by addressing stress reactivity/stress resilience, the psychological and physiological response of the body to stress, as the underlying mechanism to facilitate behavioral change. In this way the study can improve health outcomes (caregiver stress, quality of life, cardiovascular disease risk).

DETAILED DESCRIPTION:
More than 60% of all informal Alzheimer's disease and related dementias caregiving costs are borne by African American women. Not only do these women face the known deleterious effects from caregiving stress, but also the deleterious effects from hypertension: reduced quality of life and longevity, disability, cognitive decline, and strokes. Indeed, the cumulative index of hypertension by age 55 is 75.7% for African American women compared to 40% for White women. Despite the prevalence of hypertension among African American women, to the investigator's knowledge, there are no interventions that target the complexity of chronic caregiving stress and hypertension self-care for African American women caregivers. The purpose of this pilot two-group randomized controlled pilot (N=28) is to determine the feasibility and acceptability of Mindfulness in Motion (MIM) plus the Dietary Approaches to Stop Hypertension (DASH) compared to an attention control group (Alzheimer's Association Care Training Resources) in African American caregivers with hypertension. MIM includes mindful awareness and movement from chair/standing positions, breathing exercises, healthy sleep, and guided mindfulness meditation. DASH (tailored for African Americans) uses a critical thinking approach that involves problem solving, participant-centered goal setting, health coaching, reflection, and development of self-efficacy (confidence) to promote physical activity and healthy eating. The attention control, Care Training consists of healthy living for participant's brain and body and effective communication. Randomized participants will receive the MIM DASH or Caregiver Training in 8 weekly 1-hour group sessions via telehealth. Both groups will receive bi-monthly coaching calls after completion of the 8-week intervention for 2-months. The central hypothesis is that by addressing caregiving stress reactivity/stress resilience, as the underlying mechanism to facilitate behavioral change, the intervention will also be successful in enhancing hypertension self-care. Study aims are to: (1) Determine the feasibility and acceptability of MIM DASH and Caregiver Training for African American women caregivers (age 40 and older) with hypertension; (2) Explore the impact of MIM DASH as compared to Caregiving Training control on caregiver stress (primary) and systolic blood pressure (secondary); and (3) Examine caregiver stress reactivity/stress resilience as the potential mechanism of action between the MIM DASH intervention and behavior change. Feasibility and acceptability data (e.g., screening to enrollment and treatment-specific preference ratings) will be collected throughout the study. Perceived stress, hair cortisol, stress resilience/stress reactivity, systolic blood pressure, self-care practice (stress management, nutrition, and physical activity) data are collected at baseline, 3-months, 3-months, and 9-months. This pilot will make a substantive contribution to the science of behavior change by identifying basic mechanisms, in the adoption of healthy behaviors, which can be used to implement self-care interventions to reduce health disparities in African Americans. Findings from the pilot study will inform the infrastructure for an R01 to the National Institutes on Aging.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of Hypertension (HTN) treated with an antihypertensive medication;
* age 40 and older
* a caregiver rating of the People Living With Dementia (PLWD) of 2 or greater on the Alzheimer's Dementia-8 scale;
* caregiver provides unpaid care to a PLWD at least 10 hours per week or assists with at least one instrumental activity of daily living
* self-identifies as Black/African American;
* English speaking; and
* access to a telecommunications device such as the internet via desktop, laptop/tablet, smartphone, or telephone.

Exclusion criteria:

* expect to move out of the area within 9 months;
* diagnosis of resistant HTN (blood pressure that remains above goal despite concurrent use of a diuretic/water pill and at least two other antihypertensive agents of different classes); or
* active participation in mindfulness/yoga program. The National Institute of Aging Common Data Screening and Enrollment forms will be used to track data.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Wright, PhD, Principal Investigator — Ohio State University
Locations (1):
- College of Nursing Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be disseminated using multiple strategies, such as making our results available to the NIH ClinicalTrials.gov website, transmitting them to the aging research community through peer-reviewed journals, and giving presentations of the results of the study at national and international scientific meetings. Additionally, presentations will be given to the local African American community to churches, Alzheimer's disease support groups, and beauty salons.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data will not be shared due to the regulation not pertaining to this grant
Access Criteria: Individual participant data will not be shared due to the regulation not pertaining to this grant

REFERENCES:
- [Derived] Wright KD, Richards Adams IK, Helsabeck NP, Rose KM, Moss KO, Nemati D, Palmer N, Kim B, Pokhrel Bhattarai S, Nguyen C, Addison D, Klatt MD. Stress and Hypertension Among African American Female Family Caregivers of Persons Living With Alzheimer Disease and Related Dementias: Protocol for a Pilot Internet-Based Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 27;14:e66975. doi: 10.2196/66975. PMID 40146982

RESULTS

PARTICIPANT FLOW:
Groups:
- MIM-DASH: A trained MIM provider and dietitian will deliver the MIM DASH group intervention in eight weekly 1-hour sessions via telehealth.
  Caregiver Training: A trained MIM provider and dietitian will deliver the MIM DASH group intervention in eight weekly 1-hour sessions via telehealth. Participants will receive session materials so they can follow along. Each MIM session consists of material related to mindfulness-the somatic mind/body connection, relaxation, yoga, meditation, self-awareness, and bodily cues relating to emotional reactivity. Group interaction centers on sharing ideas toward effective practice and practical daily challenges to being mindful. Each class begins with a prompt for participant contemplation during the next hour that reference a unique weekly theme which will be reiterated in the session materials.
  The DASH portion, led by the Registered Dietitian, focuses on education to increase vegetables, fruits, whole grains and decrease intakes of fat and sodium, sugar sweetened beverages and sweets. Education includes adapting traditional "Soul" food dishes to meet the DASH dietary guidelines.
Period: Overall Study
Arm/Group | MIM-DASH | Attention Control
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MIM-DASH | Attention Control | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 61.9 (7.52) | 62.9 (8.67) | 62.4 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 13 | 25
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Employment Status [Count of Participants; unit: Participants]
  Full-Time Employment | 6 | 10 | 16
  Part-Time Employment | 1 | 0 | 1
  Retired | 5 | 2 | 7
  Not Employed | 1 | 0 | 1
  Unknown/Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure (Systolic)
Description: Change is being assessed in systolic blood pressure measured with an automatic blood pressure cuff. Results outside of the normal range (90/60 to 120/80 mmHg), both higher and lower are considered undesirable.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
mmHg
  Baseline | 129 (18) | 127 (20)
  3 month | 122 (16) | 124 (17)
  9 month | 132 (12) | 122 (17)

2. Primary Outcome: Change in Blood Pressure (Diastolic)
Description: Change is being assessed in diastolic blood pressure measured with an automatic blood pressure cuff. Results outside of the normal range (90/60 to 120/80 mmHg), both higher and lower are considered undesirable.
Time Frame: Baseline, 3 month, 9 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
mmHg
  Baseline | 77 (8) | 82 (11)
  3 month | 72 (10) | 76 (11)
  9 month | 80 (10) | 76 (8)

3. Primary Outcome: Change in Heart Rate
Description: Change in heart rate is being assessed with an automatic blood pressure cuff. Results outside of the normal range (60 to 100 beats per minute), both higher and lower, are considered undesirable.
Time Frame: Baseline, 3 month, 9 month
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
Beats per minute
  Baseline | 73 (15) | 71 (7)
  3 month | 77 (12) | 71 (13)
  9 month | 70 (10) | 73 (11)

4. Secondary Outcome: Newest Vital Sign
Description: Measure of health literacy. Scores range from 0-6 with lower scores indicating lower health literacy
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale | 4.23 (1.69) | 3.92 (1.71)

5. Secondary Outcome: Change is Being Assessed in Stress Management Practices Survey Part A
Description: A list of 13 statements such as "I am able to use muscle relaxation techniques to reduce any tension I experience" that is measured on a Likert scale. Scores range from 0 to 52 with higher scores indicating greater use of stress management strategies.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 34.54 (9.13) | 40.46 (7.11)
  3 month | 39.31 (6.58) | 38.2 (7.47)
  9 mon th | 35.93 (8.76) | 35.92 (6.26)

6. Secondary Outcome: Change is Being Assessed in Perceived Stress Scale (Caregiver Stress)
Description: The Perceived Stress Scale has 10-items one a Likert scale with a reference range of 0-30 regarding stress over the past month. Values are: 0 - Never, 1 - Almost Never, 2 - Sometimes, 3 - Fairly Often, 4 - Very Often The investigators will sum 10 items to create a composite score, ranging from 0 to 40.
  The higher score, the higher levels of perceived stress.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 14.93 (7.27) | 14.57 (6.36)
  3 month | 14.92 (6.5) | 10.78 (3.73)
  9 month | 12.57 (7.85) | 10.75 (5.82)

7. Secondary Outcome: Change is Being Assessed in in World Health Organization Quality of Life (WHO-5 QOL)
Description: The World Health Organization (WHO-5) is a short questionnaire consisting of five Likert scale statements of well-being over the past 2-weeks. Scores range from 0-25. Higher scores represent higher quality of life
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 13.79 (5.91) | 16.83 (3.46)
  3 month | 13.83 (5.13) | 17.67 (2.65)
  9 month | 15.14 (5.53) | 16.2 (3.29)

8. Secondary Outcome: Change is Being Assessed in Generalized Anxiety Symptom Scale
Description: Generalized Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). The GAD-7 represents an anxiety measure based on seven items which are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 5.64 (4.07) | 3.29 (2.89)
  3 month | 4.46 (3.93) | 3.8 (2.82)
  9 month | 3.5 (3.7) | 2.33 (2.06)

9. Secondary Outcome: Change is Being Assessed in Revised Memory and Behavior Checklist
Description: Assess psychological comorbidity of the caregiver and health status of the person living with ADRD. 32-item check-list that assess activities of daily living and problem behaviors in people living with Alzheimer's disease and related dementias (AD/ADRD). Scores range from 0-96 with higher indicating more behavioral problems in the care recipient
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 20.57 (15.34) | 15.92 (11.43)
  3 month | 18.58 (12.43) | 15.5 (11.3)
  9 month | 14 (10.17) | 16.3 (13.94)

10. Secondary Outcome: Credibility Scale
Description: The Credibility Scale measures attitudes towards the treatment condition and the participants' expectation of benefit once the treatment has been explained. The scale consists of 5 questions rated on a 0 (not at all confident) to 10 (very confident). The range of scores is from 0 - 50. Higher scores, up to 45, will indicate greater credibility of the treatment condition.
  There are no subscales in this tool.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale | 41.23 (4.92) | 41.42 (3.37)

11. Secondary Outcome: Acceptability Scale
Description: Treatment-specific preference ratings (pre- and post-intervention).The participants will complete the Acceptability of Participant Preferences 13-item Likert-type survey ranging from 1 (strongly disagree) to 5 (strongly agree). Scores can range from 13 - 65. Higher scores indicate that participants find the intervention more acceptable.
  There are no subscales in this tool.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale | 59.08 (7.38) | 60.83 (5.56)

12. Secondary Outcome: Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4)
Description: The K-Wood-MAS-4 is a self-report 4-item, hybrid tool developed to capture four domains of adherence behavior: self-efficacy, physical function, intentional medication-taking, and forgetfulness. The 4-item scale categorizes participants as low and high adherence. Scores range from 0 to 4 with a score of 1 or greater indicating lower prescription medication adherence.
  There are no sub-scales in this tool.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 1.214 (1.188) | 1.077 (1.115)
  3 month | 1.167 (1.267) | 1 (1.247)
  9 month | 0.929 (0.917) | 1.091 (1.221)

13. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a 9-item measure of depression and each item is scored on a scale of 0-3. The total ranges from 0-27 (scores of 5-9 are mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; and 20 severe depression). Higher scores indicate worse depression and worse outcomes.
  There are no subscales in this tool.
Time Frame: Baseline, 3 months, 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MIM-DASH | Attention Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Baseline | 4.86 (3.61) | 3.69 (2.72)
  3 month | 6.23 (4.82) | 3.9 (2.47)
  9 month | 3.62 (3.36) | 3.42 (2.35)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during the 8 week intervention period, and throughout the follow up period of up to 9 months.
Description: Adverse Event definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | MIM-DASH | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05721482/Prot_SAP_002.pdf
  • Informed Consent Form (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT05721482/ICF_003.pdf